CLINICAL TRIAL: NCT02556411
Title: Comparison of E/P Therapy in Continuous Regimen Versus Combination of LNG-IUS Plus E/P
Brief Title: Comparison of Estrogen-progestin Therapy in Continuous Regimen Versus Combination Estrogen-progestin Therapy in Continuous Regimen Plus Levonorgestrel-releasing Intrauterine System (LNG-IUS)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Cagliari (Other)
Responsible Party: Principal Investigator, Stefano Angioni, Associate Professor, University of Cagliari
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADENOMYOSIS
Record Dates: First submitted 2015-09-20; First posted 2015-09-22 (Estimated); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Adenomyosis; Chronic Pelvic Pain
MeSH Terms: conditions — Adenomyosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LNG-IUS (Active Comparator): LNG-IUS 13,5 mg di Levonorgestrel
  Interventions: Drug: LNG-IUS 13,5 mg Levonorgestrel
- combined oral contraceptive plus LNG-IUS (Experimental): Levonorgestrel 0,10 mg+ ethinylestradiol 0,02 mg+ LNG-IUS 13,5 mg di Levonorgestrel
  Interventions: Drug: LNG-IUS 13,5 mg Levonorgestrel; Drug: Levonorgestrel 0,10 mg+ ethinylestradiol 0,02 mg

INTERVENTIONS:
Drug: LNG-IUS 13,5 mg Levonorgestrel — LNG-IUS
Drug: Levonorgestrel 0,10 mg+ ethinylestradiol 0,02 mg — Levonorgestrel 0,10 mg+ethinylestradiol 0,02 mg oral contraceptive pill in continuous regime
  Arms: combined oral contraceptive plus LNG-IUS

SUMMARY:
Adenomyosis is characterized by the appearance of endometrial cells in the muscular layer of the uterus. It affects about 15-20% of the female population.

The symptoms of adenomyosis are heavy menstrual bleedings and painful menstruation (dysmenorrhea) and in addition chronic pelvic pain. Regarding treatment levonogestrel-releasing intrauterine system, Gonadotropin releasing hormone (GnRH)-analogues, Danazol, uterine embolization and endometrial ablation have been tried. The aim of this study is to compare the efficacy and usefulness of association of oral contraceptive pill and LNG-IUS or LNG-IUS alone

ELIGIBILITY:
Inclusion Criteria:

* Women affected by adenomyosis with pelvic pain > 4;
* Negative Pap Smear test

Exclusion Criteria:

* Pregnancy or research of pregnancy
* Refusal or inability to sign informed consent
* Severe underlying comorbidities (hepatic, oncological)
* Pelvic inflammatory disease
* Other cervical or uterine pathologies
* Deep venous thromboembolism
* Hormonal therapy contraindications
* Smoke

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Change of Pelvic pain as measured by visual analogue scale | Change from baseline pelvic pain at 45 days of treatment

SECONDARY OUTCOMES:
Change of Pelvic pain as measured by visual analogue scale | Change from baseline pelvic pain at 90 days of treatment
Change of Pelvic pain as measured by visual analogue scale | Change from baseline pelvic pain at 180 days of treatment
Change of Pelvic pain as measured by visual analogue scale | Change from baseline pelvic pain at 365 days of treatment
Quality of sexual life | Cases were administered and fulfilled the questionnaires at the moment of diagnosis of adenomyosis up to 4weeks; Change from baseline were evaluated 45 days after begin of treatment